CLINICAL TRIAL: NCT03490201
Title: FLExAbility Sensor Enabled Substrate Targeted Ablation for the Reduction of Ventricular Tachycardia (LESS-VT) Study
Brief Title: FLExAbility Sensor Enabled Substrate Targeted Ablation for the Reduction of VT Study
Acronym: LESS-VT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SJM-CIP-10138
Record Dates: First submitted 2017-08-28; First posted 2018-04-06 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: Pivotal medical device study
Who Masked: Participant
Masking Description: Subjects are blinded to the randomization assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Randomized - Control (Active Comparator): Subjects with ICM and randomized to the Control group will undergo mapping and substrate-based ablation for the treatment of ventricular tachycardia with any of the protocol-specified commercially available ablation catheters indicated for patients with ICM. A protocol-specified commercially available mapping system will be used in conjunction with the control catheter in the ablation procedure. Subjects will be followed for 12 months post-procedure.
  Interventions: Device: Market Approved RF Ablation System
- Randomized - Treatment (Active Comparator): Subjects with ICM and randomized to the Treatment group will undergo mapping and substrate-based ablation for the treatment of ventricular tachycardia with the investigational FlexAbility SE Catheter. The Ampere Generator, Cool Point Irrigation Pump and the EnSite Precision Cardiac Mapping System or EnSite X EP System will be used in conjunction with the FlexAbility SE catheter in the ablation procedure. Subjects will be followed for 12 months post-procedure.
  Interventions: Device: FlexAbility SE Ablation Catheter
- Non-randomized - Treatment (Experimental): Subjects with NICM will undergo mapping and substrate-based ablation for the treatment of ventricular tachycardia with the investigational FlexAbility SE Catheter. The Ampere Generator, Cool Point Irrigation Pump and the EnSite Precision Cardiac Mapping System or EnSite X EP System will be used in conjunction with the FlexAbility SE catheter in the ablation procedure. Subjects will be followed for 12 months post-procedure.
  Interventions: Device: FlexAbility SE Ablation Catheter

INTERVENTIONS:
Device: Market Approved RF Ablation System — Subjects receive ablation using an FDA approved radiofrequency (RF) ablation system.
  Arms: Randomized - Control
Device: FlexAbility SE Ablation Catheter — Subjects receive ablation treatment using an ablation system that is not FDA approved.
  Arms: Non-randomized - Treatment; Randomized - Treatment

SUMMARY:
This clinical investigation is intended to demonstrate the safety and effectiveness of ventricular ablation therapy using the FlexAbility Sensor Enabled Ablation Catheter in patients with drug-refractory monomorphic ventricular tachycardia in whom ventricular tachycardia recurs despite antiarrhythmic drug therapy or when antiarrhythmic drugs are not tolerated or desired.

DETAILED DESCRIPTION:
This is a regulated, prospective, multi-center trial designed to evaluate the safety and effectiveness of the FlexAbility[TM] Ablation Catheter, Sensor Enabled[TM] (FlexAbility SE) catheter to obtain an indication to treat monomorphic ventricular tachycardia (MMVT) in the United States of America (US). The clinical trial has two cohorts: one is a randomized ischemic cardiomyopathy (ICM) cohort and the second is a concurrent single-arm non-ischemic cardiomyopathy (NICM) cohort. Four hundred ten (410) subjects with drug refractory sustained MMVT and ICM and 182 subjects with drug refractory sustained MMVT and NICM will be enrolled at up to 35 centers worldwide. Study subjects who have drug refractory sustained MMVT and ICM will be randomized 1:1 to treatment with the FlexAbility SE catheter ablation system in the Treatment group, or the ThermoCool, ThermoCool NaviStar, or ThermoCool SmartTouch Ablation Catheter from Biosense Webster in the Control group. Since at study start there was no approved device for VT ablation in patients with NICM to use as a comparator, subjects who have drug refractory MMVT and NICM will be treated with the FlexAbility SE catheter ablation system only.

ELIGIBILITY:
Inclusion Criteria:

* Structural heart disease (ischemic or non-ischemic) with one of the following:

  * Confirmed diagnosis via echocardiography and/or cardiac CT/MRI [computed tomography/magnetic resonance imaging], or
  * Left ventricular ejection fraction (EF) <40% (documented within the last 6 months via echocardiography, or
  * Arrhythmogenic RV [right ventricular] cardiomyopathy/dysplasia (per 2010 ARVC/D [arrhythmogenic right ventricular cardiomyopathy/dysplasia] Task Force Criteria).27
* At least one documented episode of sustained MMVT by either EGM [cardiac electrogram] or ECG [electrocardiogram] in the 6 months prior to enrollment
* Implanted with a market released ICD [implantable cardioverter-defibrillator] or CRT-D [cardiac resynchronization therapy-defibrillator] for at least 30 days prior to index ablation procedure
* Refractory (i.e. not effective, not tolerated or not desired) to at least one anti-arrhythmic medication (either amiodarone or sotalol) for treatment of MMVT
* At least 18 years of age
* Informed of the nature of the study, agreed to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee (IRB/EC) of the respective clinical study site.
* Able and willing to comply with all study requirements

Exclusion Criteria:

* Implanted with a subcutaneous ICD
* Implanted with a ventricular assist device (VAD) (e.g. TandemHeart)
* Currently receiving support, or anticipated to receive support prior to the index ablation procedure, via extracorporeal membrane oxygenation (ECMO)
* Presence of intracardiac thrombus verified via computer tomography (CT), magnetic resonance imaging (MRI), transesophageal echocardiogram (TEE), or transthoracic echocardiogram (TTE) within 48 hours prior to the index ablation procedure or intra-procedure intracardiac echocardiography (ICE)

  o For subjects with a history of AF [atrial fibrillation], this verification must be done via TEE or ICE
* ST elevation myocardial infarction (MI) within 60 days prior to index ablation procedure
* Previous cardiac surgery (e.g. ventriculotomy, atriotomy, coronary artery bypass graft), within 60 days prior to index ablation procedure
* Percutaneous coronary intervention (PCI) within 30 days prior to index ablation procedure
* Idiopathic VT
* Incessant VT (continuous sustained VT that promptly recurs despite repeated intervention for termination over ≥3 hours) necessitating immediate treatment or requiring hemodynamic support prior to the ablation procedure
* VT/VF [ventricular tachycardia/ventricular fibrillation] thought to be from channelopathies
* Reversible cause of VT
* Severe aortic stenosis or flail mitral valve
* Mechanical mitral and aortic valve
* History of stroke with modified Rankin scale > 3 (See Appendix C)
* Unstable angina
* Chronic NYHA [New York Heart Association] Class IV heart failure
* Ejection fraction < 15%
* Thrombocytopenia (defined as platelet count <80,000) or coagulopathy
* Contraindication to systemic anticoagulation (i.e. heparin, warfarin, or a direct thrombin inhibitor)
* Women who are pregnant or nursing
* Active uncontrolled infection
* Other anatomic or co morbid conditions or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the patient's ability to participate in the study or to comply with follow up requirements, or impact the scientific soundness of the study results
* Enrolled in an investigational study evaluating another device or drug that would confound the results of this study
* Have a life expectancy of less than 12 months due to any condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Rate of complications | 7 days
  The primary safety endpoint is a composite of cardiovascular-related and procedure-related major complications through 7 days post index ablation procedure.
Freedom from recurrence of VT | 6 months
  The primary effectiveness endpoint is freedom from recurrent sustained MMVT at 6 months and a new or increased dose Class I or III antiarrhythmic drugs (AAD) at 6 months following the index ablation procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kammer, Study Director — Abbott
Locations (32):
- United States (23):
  - Affinity Cardiovascular Specialists, LLC, Birmingham, Alabama
  - University Hospital - Univ. of Alabama at Birmingham (UAB), Birmingham, Alabama
  - USC University Hospital, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of California at San Diego (UCSD) Medical Center, San Diego, California
  - University of Colorado Hospital, Aurora, Colorado
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - University of South Florida, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - VA Medical Center Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - WakeMed Hospital, Raleigh, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Heart and Vascular Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia, Austin, Texas
  - Texas Heart Institute, Houston, Texas
  - Memorial Hermann Hospital, The Woodlands, Texas
  - University of Washington, Seattle, Washington
- Royal Adelaide Hospital, Adelaide, South Australia, Australia
- Czechia (2):
  - IKEM, Prague, Central Bohemia
  - Nemocnice Na Homolce, Prague
- Hopital Haut Leveque, Pessac, France
- Herzzentrum Leipzig GmbH, Leipzig, Germany
- Italy (2):
  - Ospedale San Raffaele, Milan
  - Centro Cardiologico Monzino, Milan
- Hospital General Universitario Gregorio Marañón, Madrid, Spain
- St. Georges Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No